CLINICAL TRIAL: NCT03938103
Title: A Hybrid Effectiveness-implementation Trial of Go NAPSACC: A Childcare-based Obesity Prevention Program
Brief Title: Evaluation of an Enhanced Delivery Model for Go NAPSACC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of Kentucky (Other); Child Care Aware of Kentucky (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 19-0406; R01HL137929 (NIH)
Record Dates: First submitted 2019-04-29; First posted 2019-05-06 (Actual); Results first posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2022-10

CONDITIONS: Obesity
Keywords: preschool; child care centers; nutrition; physical activity; organizational readiness; behavior change; cost-effectiveness; implementation
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Go NAPSACC (Experimental): Enhanced delivery model
  Interventions: Behavioral: Enhanced Go NAPSACC
- Basic Go NAPSACC (Active Comparator): Basic delivery model
  Interventions: Behavioral: Basic Go NAPSACC

INTERVENTIONS:
Behavioral: Enhanced Go NAPSACC — In the Enhanced delivery model, TA coaches will help centers create an implementation team and conduct a needs assessment to identify organizational strengths and challenges. TA coaches will also provide an orientation to Go NAPSACC and its online tools and help the team develop a plan to guide their Go NAPSACC efforts. The team will then work through 2 cycles of Go NAPSACC over 12 months. During each cycle (6 months), centers will take self-assessments on nutrition and physical activity, choose 6 goals (3 from each), create action plans, and take action to achieve their chosen goals. Throughout this 12-month period, TA coaches will provide monthly check-ins incorporating tailored support based on the results from the needs assessment. They will also organize 2-3 meetings among teams from different centers to reflect and share lessons learned.
  Arms: Enhanced Go NAPSACC
Behavioral: Basic Go NAPSACC — In the Basic delivery model, TA coaches will provide an orientation to Go NAPSACC and its online tools to the center director. The director will then work 2 cycles of Go NAPSACC over 12 months. During each cycle (6 months), centers will take self-assessments on nutrition and physical activity, choose 6 goals (3 from each), create action plans, and take action to achieve their chosen goals. Throughout this 12-month period, TA coaches will provide monthly brief check-ins.
  Arms: Basic Go NAPSACC

SUMMARY:
This study will compare the effectiveness and cost of Basic and Enhanced delivery models for Go NAPSACC on child care centers' use of evidence-based nutrition and physical activity practices. Technical assistance (TA) coaches from Child Care Aware of Kentucky will lead delivery. Half of the TA coaches will deliver Go NAPSACC using the Basic model and the other half will deliver the program using the Enhanced model. It is hypothesized that the Enhanced model will result in greater use of evidence-based nutrition and physical activity practices and will also be more cost effective.

DETAILED DESCRIPTION:
This research study will use a type 3 hybrid effectiveness-implementation design with a randomized controlled trial to evaluate the impact of Go NAPSACC when using basic vs enhanced implementation models (i.e., Basic Go NAPSACC vs. Enhanced Go NAPSACC). To evaluate impact, measures collected at baseline and post-intervention will be used to assess change in centers' use of evidence-based nutrition and physical activity practices. Cost of delivery will also be monitored throughout implementation. Study participants will include 28 TA coaches from Child Care Aware of Kentucky and 97 child care centers from 7 regions of central Kentucky.

ORIGINAL RECRUITMENT: First, TA coaches will attend an orientation session where they will be introduced to the research study and their roles both as study participants and implementation partners. If they agree to participate, they will be asked to sign consent. TA coaches will then be trained on how to introduce the research study to child care centers using provided recruitment materials. They will be instructed to target these efforts toward a randomly selected list of centers (drawn from their current caseload) provided by the research team. Coaches will be responsible for gauging initial interest of centers, and relaying that information to the research team. Research staff will follow up directly with all centers who express initial interest to confirm eligibility and interest, review study details, and answer questions. Once a center director's eligibility and interest is confirmed, the research team will work with the director to recruit a randomly selected 3-4-year-old classroom teacher and at least three 3-4-year-old children from that classroom.

RELAUNCH RECRUITMENT: TA coaches will attend a re-orientation session where they will be informed of modifications to the study due to the pandemic restrictions. For the first two waves, TA coaches will be instructed to inform their previously enrolled centers of the modifications to the study. They will be provided with materials to inform centers and relay any relevant information about their centers to the research staff. Research staff will follow-up directly with all previously enrolled centers who are currently open. The research study staff will review study details, confirm interest, and answer any questions. Once a center director's interest is confirmed, the staff will work with the director to recruit two randomly selected preschool classroom teachers. Wave 3 TA coaches will be informed of modifications to study and follow a similar protocol to the original recruitment steps as measurement wasn't complete at the time of the pause due to the pandemic. The TA coaches will use provided recruitment materials and will be instructed to target these efforts toward a randomly selected list of centers (drawn from their current caseload) provided by the research team. Coaches will be responsible for gauging initial interest of centers, and relaying that information to the research team. Research staff will follow up directly with all centers who express initial interest to confirm eligibility and interest, review study details, and answer questions. Once a center director's eligibility and interest is confirmed, the research team will work with the director to recruit two randomly selected preschool classroom teachers.

ORIGINAL BASELINE MEASURES: Several measures will be collected at baseline on centers, children, directors, teachers, and TA coaches using a combination of observation, physical assessments, and self-report surveys. Most measures will be collected during a 1-day site visit conducted with each center by a trained research team member. Measures will assess centers' use of evidence-based nutrition and physical activity practices, children's dietary intakes and physical activity while at child care, and children's height and weight. Demographic information will be captured through surveys completed by parents, directors, teachers, and TA coaches. Implementation context will be captured through surveys completed by directors, teachers, and TA coaches.

RELAUNCH BASELINE MEASURES: Several measures will be collected at baseline on centers, directors, teachers and TA coaches using online self-report surveys. All measures will be collected using the Qualtrics online survey tool. For TA coaches, measures will assess demographics information, implementation context, and COVID-19 impact. For center directors, measures will assess demographics, center demographics, implementation context, COVID-19 impact, and nutrition and physical activity practices. For preschool teachers, measures will assess demographics, implementation context, and nutrition and physical activity practices.

RANDOMIZATION: Once all baseline measures with centers are scheduled, TA coaches will be randomly assigned to either deliver Basic or Enhanced Go NAPSACC with their enrolled centers. For Wave 3, once all online baseline measures are completed, TA coaches will be randomly assigned to either deliver Basic or Enhanced Go NAPSACC with their enrolled centers.

INTERVENTION ARMS: Go NAPSACC is a suite of online tools designed to help child care programs improve their nutrition and physical activity practices. TA coaches will support centers' use of Go NAPSACC using either a Basic or Enhanced implementation model.

TA coaches assigned to Basic Go NAPSACC will participate in 2 two hour-long training sessions and a homework assignment. Training sessions will cover the role of child care programs in shaping children's eating and physical activity behaviors, Go NAPSACC's 5-step improvement, and the tools available for child care programs and TA coaches to support their work. Additionally, coaches will have an online check-in meeting 1 month post-training to answer any remaining questions/concerns. TA coaches assigned to Enhanced Go NAPSACC will participate in 2 two hour long and 2 hour-long training sessions and a homework assignment. In addition to the topics listed above, trainings will also introduce elements unique to the enhanced implementation model. During implementation, these TA coaches will also participate in monthly conference calls and 2-3 one-on-one coaching sessions with a Go NAPSACC specialist .

For centers receiving Basic Go NAPSACC, center directors will be invited by their TA coach to register for Go NAPSACC accounts. The director will receive a 1-hour orientation from their TA coach on how to use Go NAPSACC's online tools and resources. Once trained, the director will complete 2 cycles of Go NAPSACC's 5-step improvement process focusing on child nutrition and physical activity. A cycle of Go NAPSACC includes completing nutrition and physical activity self-assessments, choosing at least 6 goals (3 goals per self-assessment), creating an action plan for each goal, working to implement the action plans drawing from the tips and materials resource library, and logging progress and completion of goals. Each cycle will take approximately 6 months to complete. At the end of the 12 months, the director will retake the self-assessments on child nutrition and physical activity. Throughout the 12 months, the director will receive brief monthly check-ins from their TA coach. TA coaches will log their implementation activities using the TA Activity Log in Go NAPSACC.

For centers receiving Enhanced Go NAPSACC, center directors will work with their TA coach to identify an implementation team that will contribute to Go NAPSACC efforts. Before starting Go NAPSACC, the team will work with their TA coach to conduct an assessment of their center's needs, capacity, and resources. A needs assessment survey will be completed by various center staff and scored by the TA coach. Summarized results will be presented and discussed with the team to identify priority issues the team would like extra support from the TA coach as they work through Go NAPSACC. Once this needs assessment is complete, the team will begin using Go NAPSACC and with support from their TA coach will create a 12-month plan to guide their Go NAPSACC efforts. Similar to those assigned to Basic Go NAPSACC, the team will complete 2 cycles of the 5-step improvement process focusing on nutrition and physical activity. They will follow the same steps described above. Additionally, the team will receive brief check-ins with tailored support from their TA coach. Further, their TA coach will host 2-3 one-hour meetings with different centers from the same region so that teams can reflect on their efforts and share lessons learned. TA coaches will be asked to log all of their implementation activities using the TA Activity Log in Go NAPSACC.

REFRESHER INTERVENTION TRAINING SESSIONS: For Waves 1 and 2, Basic TA coaches will have 2 hour and a half long online refresher training sessions. The first training session will cover a refresher on the 5-step process, the provider and consultant online tools, and timeline updates. The second session will focus on providing support remotely and on how Go NAPSACC best practices may be impacted by pandemic restrictions. Enhanced coaches will have a 2-hour training session focused on a reminder of the big picture of the Enhanced support approach, the updated timeline, leadership team formation, the readiness check, and providing support remotely. Regular monthly meetings will be used to further refresh on topics relevant to Enhanced support approach and how best practices could be impacted by pandemic restrictions.

POST-INTERVENTION MEASURES: Measures will be repeated following 12 months of Go NAPSACC participation. Data collection procedures will be the same as those described in relaunch baseline measures. In addition, trained research staff will complete phone interviews with a random selection of TA coaches to gather feedback about their experiences implementing Go NAPSACC. Phone interviews will also be completed with randomly selected center directors and when relevant, members of the implementation teams.

ELIGIBILITY:
Inclusion Criteria:

TA Coaches

* Must either be a Quality coach or a Health and Safety coach
* Must be able to read and speak English

Child Care Centers

* Must be a part of a participating TA coach's current caseload
* Have no plans to close in the coming year
* Serve at least lunch to the children
* Not serve special needs children exclusively

Child Care Providers

* Teacher must be the lead teacher in a preschool classroom
* Center directors and teachers must be able to read and speak English

Exclusion Criteria:

Child Care Centers

* Serve special needs children exclusively
* Serve only non-English speaking families

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 364 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2022-10-07 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dianne Ward, EdD, Principal Investigator — University of North Carolina, Chapel Hill; Derek Hales, PhD, Principal Investigator — University of North Carollina at Chapel Hill
Locations (2):
- United States (2):
  - University of Kentucky, Lexington, Kentucky
  - UNC Chapel Hill, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Time Frame: Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication.
Access Criteria: The investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.

REFERENCES:
- [Background] Fernandez ME, Walker TJ, Weiner BJ, Calo WA, Liang S, Risendal B, Friedman DB, Tu SP, Williams RS, Jacobs S, Herrmann AK, Kegler MC. Developing measures to assess constructs from the Inner Setting domain of the Consolidated Framework for Implementation Research. Implement Sci. 2018 Mar 27;13(1):52. doi: 10.1186/s13012-018-0736-7. PMID 29587804
- [Background] Lehman WE, Simpson DD, Knight DK, Flynn PM. Integration of treatment innovation planning and implementation: strategic process models and organizational challenges. Psychol Addict Behav. 2011 Jun;25(2):252-61. doi: 10.1037/a0022682. PMID 21443294
- [Background] Seward K, Wolfenden L, Wiggers J, Finch M, Wyse R, Oldmeadow C, Presseau J, Clinton-McHarg T, Yoong SL. Measuring implementation behaviour of menu guidelines in the childcare setting: confirmatory factor analysis of a theoretical domains framework questionnaire (TDFQ). Int J Behav Nutr Phys Act. 2017 Apr 4;14(1):45. doi: 10.1186/s12966-017-0499-6. PMID 28376892
- [Background] Evenson KR, Catellier DJ, Gill K, Ondrak KS, McMurray RG. Calibration of two objective measures of physical activity for children. J Sports Sci. 2008 Dec;26(14):1557-65. doi: 10.1080/02640410802334196. PMID 18949660
- [Derived] Vaughn AE, Studts CR, Powell BJ, Ammerman AS, Trogdon JG, Curran GM, Hales D, Willis E, Ward DS. The impact of basic vs. enhanced Go NAPSACC on child care centers' healthy eating and physical activity practices: protocol for a type 3 hybrid effectiveness-implementation cluster-randomized trial. Implement Sci. 2019 Dec 5;14(1):101. doi: 10.1186/s13012-019-0949-4. PMID 31805973

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Childcare centers are clustered within TA coaches. TA coaches delivered part of the intervention and served as the unit of randomization. Information used to quantify aspects of each center was collected from the TA coach, directors, and staff. To clearly represent the groups of people recruited within each arm three "periods" are defined below. Periods do not reflect a time element for this study, but the three groups of people measured for center-level data (unit).
Units Other Than Participants: ChildCare Centers
Groups:
- Enhanced Go NAPSACC: Go NAPSACC implemented using enhanced delivery model, including additional coaching support, formation of leadership teams, and assessment of readiness.
- Basic Go NAPSACC: Go NAPSACC implemented using basic delivery model.
Period: Technical Assistant (TA) Coaches
Arm/Group | Enhanced Go NAPSACC | Basic Go NAPSACC
Started (TA coaches were part of intervention delivery and randomized to a study arm. "Periods" were used in this flow to represent units of people serving a childcare center.) | 14; 55 ChildCare Centers | 13; 42 ChildCare Centers
Completed | 14; 48 ChildCare Centers | 13; 39 ChildCare Centers
Not Completed | 0; 7 ChildCare Centers | 0; 3 ChildCare Centers
Period: Center Directors
Arm/Group | Enhanced Go NAPSACC | Basic Go NAPSACC
Started (Periods in this flow represent groups of child care directors recruited within centers.) | 65; 55 ChildCare Centers | 49; 42 ChildCare Centers
Completed | 48; 48 ChildCare Centers | 36; 39 ChildCare Centers
Not Completed | 17; 7 ChildCare Centers | 13; 3 ChildCare Centers
Period: Center Staff
Arm/Group | Enhanced Go NAPSACC | Basic Go NAPSACC
Started (Periods in this flow represent groups of child care staff recruited within centers.) | 128; 55 ChildCare Centers | 95; 42 ChildCare Centers
Completed | 73; 48 ChildCare Centers | 60; 39 ChildCare Centers
Not Completed | 55; 7 ChildCare Centers | 35; 3 ChildCare Centers

BASELINE CHARACTERISTICS:
Population: Demographic characteristics are summarized for all TA coaches, directors, and staff who completed surveys and provided information for center-level analysis (n=364).
Groups:
- Enhanced Go NAPSACC: Go NAPSACC implemented with the Enhanced delivery model
- Basic Go NAPSACC: Go NAPSACC implemented with the Basic delivery model
- Total: Total of all reporting groups
Arm/Group | Enhanced Go NAPSACC | Basic Go NAPSACC | Total
Number analyzed (Participants) | 207 | 157 | 364
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: missing data - participants failed to report age on questionnaire
  years
    number analyzed (Participants) | 201 | 153 | 354
    (all) | 38.69 (12.47) | 37.77 (11.81) | 38.29 (12.18)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: missing data - participants did not provide sex classification on questionnaire
  Participants
    number analyzed (Participants) | 206 | 153 | 359
    Female | 201 | 152 | 353
    Male | 5 | 1 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 10 | 13
  Not Hispanic or Latino | 199 | 141 | 340
  Unknown or Not Reported | 5 | 6 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 24 | 24 | 48
  White | 173 | 117 | 290
  More than one race | 5 | 2 | 7
  Unknown or Not Reported | 3 | 12 | 15
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 207 | 157 | 364

OUTCOME MEASURES:

1. Primary Outcome: Mean Nutrition Environment Score
Description: Each center's nutrition environment was assessed using the Environment and Policy Assessment and Observation- Self Report (EPAO-SR), a self-report measure filled out through online surveys by child care center directors and preschool classroom teachers. In addition, directors upload a month of menus and policy handbooks, which are reviewed and scored by a trained staff members. An overall nutrition environment score will be derived with scores ranging from 0-3, where higher scores indicate better (more supportive) nutrition environments.
Time Frame: Measures collected 3-12 weeks prior to start of intervention (Baseline) and 1-8 weeks post-12-month intervention (Follow-up)
Population: The unit of analysis for this outcome is center-level nutrition environment score, derived from surveys completed by directors and staff at each center. Survey responses from directors and staff must be combined to compute the nutrition environment score for a center, therefore the number of participants analyzed is the number of centers in each arm, not the total number of directors and staff.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: centers
Groups:
- Enhanced Go NAPSACC: Centers received Go NAPSACC Enhanced delivery model from TA coaches
- Basic Go NAPSACC: Centers received Go NAPSACC Basic delivery model from TA coaches.
Arm/Group | Enhanced Go NAPSACC | Basic Go NAPSACC
Number analyzed (Participants) | 193 | 144
Number analyzed (centers) | 55 | 42
score on a scale
  Baseline | 1.88 (0.24) | 1.98 (0.27)
  Follow-Up: number analyzed (Participants) | 168 | 134
  Follow-Up: number analyzed (centers) | 48 | 39
  Follow-Up | 2.06 (0.23) | 2.08 (0.26)
Statistical Analysis 1: Comparison: Enhanced Go NAPSACC vs Basic Go NAPSACC; Test type: Other; p = 0.101, Mixed Models Analysis

2. Primary Outcome: Mean Physical Activity Environment Score
Description: Each center's physical activity environment was assessed using the Environment and Policy Assessment and Observation- Self Report (EPAO-SR), a self-report measure filled out through online surveys by child care center directors and preschool classroom teachers. In addition, directors upload policy handbooks, which were reviewed by a trained staff member. An overall physical activity environment score was derived with scores ranging from 0-3, where higher scores indicate better (more supportive) physical activity environments.
Time Frame: as for outcome 1
Population: The unit of analysis for this outcome is center-level physical activity environment score, derived from surveys completed by directors and staff at each center. Survey responses from directors and staff must be combined to compute the physical activity environment score for a center, therefore the number of participants analyzed is the number of centers in each arm, not the total number of directors and staff.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: centers
Arm/Group | Enhanced Go NAPSACC | Basic Go NAPSACC
Number analyzed (Participants) | 193 | 144
Number analyzed (centers) | 55 | 42
score on a scale
  Baseline | 1.26 (0.27) | 1.33 (0.32)
  Follow-Up: number analyzed (Participants) | 168 | 134
  Follow-Up: number analyzed (centers) | 48 | 39
  Follow-Up | 1.50 (0.34) | 1.50 (0.32)
Statistical Analysis 1: Comparison: Enhanced Go NAPSACC vs Basic Go NAPSACC; Test type: Other; p = 0.383, Mixed Models Analysis

3. Secondary Outcome: Number of Centers That Created a Go NAPSACC Website Account
Description: The number of participating centers will be captured by the Go NAPSACC website and extracted using the Go NAPSACC registration report. The registration report documents all child care centers that have completed registration and created a Go NAPSACC account. Creation of an account will be used to define participation/adoption.
Time Frame: Measures collected 3-12 weeks prior to start of intervention (Baseline)
Population: Centers recruited and randomized
Measure: Count of Units; unit: Centers
Units Other Than Participants: Centers
Arm/Group | Enhanced Go NAPSACC | Basic Go NAPSACC
Number analyzed (Participants) | 55 | 42
Number analyzed (Centers) | 55 | 42
Centers | 40 | 38

4. Secondary Outcome: Go NAPSACC Core Program Components Completed by Centers
Description: Number of Go NAPSACC core program components completed was captured by the Go NAPSACC website and extracted using the Detailed Activity Report. These data serve as indicators of fidelity. The Detailed Activity report captures centers' completion of key steps in the improvement process (completion of a self-assessments and creation/completion of action plans). For this study, centers were expected to complete a cycle of the improvement process for Nutrition and one for Physical Activity, including all key steps.
Time Frame: Measures collected during the 1 year intervention period.
Population: For this outcome only childcare centers that completed registration in the Go NAPSACC website system were analyzed. As presented in outcome #3, 40 of 55 centers from the enhanced arm and 38 of 42 centers in the basic arm created an account in the Go NAPSACC website. These outcomes could only be computed for the 78 centers (40 + 38) with accounts.
Measure: Number; unit: Number of Centers
Units Other Than Participants: centers completing registration
Arm/Group | Enhanced Go NAPSACC | Basic Go NAPSACC
Number analyzed (Participants) | 40 | 38
Number analyzed (centers completing registration) | 40 | 38
Number of Centers
  Nutrition: Completed First Self-Assessment | 27 | 22
  Nutrition: Completed Second Self-Assessment | 13 | 7
  Nutrition: Completed Third Self-Assessment | 2 | 0
  Nutrition: Created Action Plan | 23 | 20
  Nutrition: Completed Action Plan | 13 | 11
  Activity: Complete First Self-Assessment | 24 | 20
  Activity: Complete Second Self-Assessment | 10 | 4
  Activity: Complete Third Self-Assessment | 2 | 0
  Activity: Created Action Plan | 21 | 14
  Activity: Completed Action plan | 11 | 5

5. Secondary Outcome: Percent of Nutrition Best Practices Met Computed From Self-assessments Completed on Go NAPSACC Website
Description: Child nutrition self-assessment scores are captured on the Go NAPSACC website when a center director completed a self-assessment at the start and end of an improvement cycle. Completing self-assessments is an intervention component that may, or may not, be used by centers. Each self-assessment item is rated on a 1-4 point scale, where higher points indicate closer compliance with best practices, with a score of 4 indicating "meets best practice". Scores are then computed as percent of best practices met (range 0 to 100%). Self-assessment data will be extracted using the Go NAPSACC Child Nutrition Self-Assessment Report pulled immediately post-intervention.
Time Frame: Within 3 months of starting intervention and again within 12 months of initiating intervention
Population: Only 49 centers (27 + 22) completed the first nutrition self-assessment. Centers without a nutrition self-assessment in the Go NAPSACC website system were not analyzed. At follow-up 13 of 27 centers from Enhanced arm and 7 of 22 centers from basic arm completed the nutrition self-assessment.
Measure: Number; unit: percentage of best practices met
Units Other Than Participants: centers completing self-assessment
Arm/Group | Enhanced Go NAPSACC | Basic Go NAPSACC
Number analyzed (Participants) | 55 | 42
Number analyzed (centers completing self-assessment) | 27 | 22
percentage of best practices met
  Baseline: number analyzed (Participants) | 27 | 22
  Baseline | 49.4 | 47.6
  Follow-up: number analyzed (Participants) | 13 | 7
  Follow-up | 63.2 | 52.4

6. Secondary Outcome: Percent of Physical Activity Best Practices Met Computed From Self-assessments Completed on Go NAPSACC Website
Description: Child physical activity self-assessment scores are captured on the Go NAPSACC website when a center completed a self-assessment at the start and end of an improvement cycle. Completing self-assessments is an intervention component that may, or may not, be used by centers. Each self-assessment item is rated on a 1-4 point scale, where higher points indicate closer compliance with best practices, with a score of 4 indicating "meets best practice". Scores are then computed as percent of best practices met (range 0 to 100%). Self-assessment data will be extracted using the Go NAPSACC Child Physical Activity Self-Assessment Report pulled immediately post-intervention.
Time Frame: Within 3 months of starting intervention and again within 12 months of initiating intervention
Population: Only 44 centers (24 + 20) completed the first physical activity self-assessment. Centers without a physical activity self-assessment in the Go NAPSACC website system are not analyzed. At follow-up 10 of 24 centers in the enhanced arm and 4 of 20 centers from the Basic arm completed the physical activity self-assessment.
Measure: Number; unit: percentage of best practices met
Units Other Than Participants: centers completing self-assessment
Arm/Group | Enhanced Go NAPSACC | Basic Go NAPSACC
Number analyzed (Participants) | 55 | 42
Number analyzed (centers completing self-assessment) | 24 | 20
percentage of best practices met
  Baseline | 31.8 | 34.4
  Follow-up: number analyzed (Participants) | 10 | 4
  Follow-up | 60.0 | 28.3

7. Secondary Outcome: Contextual Setting (Director Report) - Impact of Center Culture, Implementation Climate, Leadership Engagement, Available Resources, and Information Access at Baseline on Intervention Effects
Description: Mean total EPAO-SR scores (percent best practices met) for centers starting with high or low contextual setting support reported by directors. Director report of contextual support was assessed using baseline surveys. Specifically, Fernandez's consolidated framework for implementation research (CFIR) inner setting measure was used to assess Culture, Culture Stress, Culture Effort, Implementation Climate, Leadership Engagement, Information access, and Available Resources. Scores from theses sub-scales were averaged to create a composite "inner setting" score. To assess the impact of baseline inner setting score and intervention group on nutrition and physical activity environment best practice scores, composite "inner setting" scores were classified as high or low using a median split. This high/low indicator of contextual support was included as interaction term in analysis models (i.e. Time [baseline-followup] * Intervention Group [basic-enhanced] * Context level[high-low]).
Time Frame: as for outcome 1
Population: The unit of analysis for this outcome is center-level, derived from surveys completed by directors at each center. The sample size is the number of centers randomized to each study arm.
Measure: Mean (Standard Deviation); unit: percentage of best practices met
Units Other Than Participants: centers
Arm/Group | Enhanced Go NAPSACC | Basic Go NAPSACC
Number analyzed (Participants) | 65 | 49
Number analyzed (centers) | 55 | 42
percentage of best practices met
  Baseline: High Contextual: number analyzed (Participants) | 32 | 26
  Baseline: High Contextual: number analyzed (centers) | 27 | 22
  Baseline: High Contextual | 32.31 (7.09) | 36.94 (7.72)
  Follow-up: High Contextual: number analyzed (Participants) | 32 | 24
  Follow-up: High Contextual: number analyzed (centers) | 27 | 21
  Follow-up: High Contextual | 40.07 (10.33) | 41.47 (9.07)
  Baseline: Low Contextual: number analyzed (Participants) | 33 | 23
  Baseline: Low Contextual: number analyzed (centers) | 28 | 20
  Baseline: Low Contextual | 30.17 (8.25) | 30.11 (8.42)
  Follow-up: Low Contextual: number analyzed (Participants) | 30 | 22
  Follow-up: Low Contextual: number analyzed (centers) | 25 | 19
  Follow-up: Low Contextual | 37.20 (9.09) | 35.88 (8.66)

8. Secondary Outcome: Contextual Setting (Staff Report) - Impact of Center Culture, Implementation Climate, Leadership Engagement, Available Resources, and Information Access at Baseline on Intervention Effects
Description: Mean total EPAO-SR scores (percent best practices met) for centers starting with high or low contextual setting support reported by staff. Staff report of contextual setting support was assessed using baseline surveys. Specifically, Fernandez's consolidated framework for implementation research (CFIR) inner setting measure was used to assess Culture, Culture Stress, Culture Effort, Implementation Climate, Leadership Engagement, Information access, and Available Resources. Scores from theses sub-scales were averaged to create a composite "inner setting" score. To assess the impact of baseline inner setting score and intervention group on nutrition and physical activity environment best practice scores, composite "inner setting" scores were classified as high or low using a median split. This high/low indicator of contextual support was included as interaction term in analysis models (i.e. Time [baseline-followup] * Intervention Group [basic-enhanced] * Context level[high-low]).
Time Frame: as for outcome 1
Population: The unit of analysis for this outcome is center-level, derived from surveys completed by staff at each center. Survey responses from staff are combined to compute the contextual score for a center, therefore the number of participants analyzed is the number of centers in each arm, not the total number of staff.
Measure: Mean (Standard Deviation); unit: percentage of best practices met
Units Other Than Participants: centers
Arm/Group | Enhanced Go NAPSACC | Basic Go NAPSACC
Number analyzed (Participants) | 128 | 95
Number analyzed (centers) | 55 | 42
percentage of best practices met
  Baseline: High Contextual: number analyzed (Participants) | 61 | 50
  Baseline: High Contextual: number analyzed (centers) | 26 | 22
  Baseline: High Contextual | 31.74 (8.35) | 34.13 (8.58)
  Follow-up: High Contextual: number analyzed (Participants) | 58 | 47
  Follow-up: High Contextual: number analyzed (centers) | 25 | 21
  Follow-up: High Contextual | 37.56 (10.12) | 39.63 (10.63)
  Baseline: Low Contextual: number analyzed (Participants) | 67 | 43
  Baseline: Low Contextual: number analyzed (centers) | 29 | 19
  Baseline: Low Contextual | 30.75 (7.19) | 34.15 (8.11)
  Follow-up: Low Contextual: number analyzed (Participants) | 63 | 41
  Follow-up: Low Contextual: number analyzed (centers) | 27 | 18
  Follow-up: Low Contextual | 39.74 (9.49) | 37.96 (7.72)

9. Secondary Outcome: Cost of Implementation for Enhanced and Basic Models
Description: Costs of implementation per center include TA coaches time and any resources required to train and support centers for 12 months. Cost tracking used the TA Activity Log to capture TA coaches' time and a supplemental log of additional costs (e.g., mileage, printing). These data were combined to calculate the average cost per center for implementing Go NAPSACC. Final amounts are expressed as cost (dollar $) per center.
Time Frame: Measures collected throughout the 1 year intervention period
Population: The sample size is the number of centers randomized to each study arm.
Measure: Mean (Standard Deviation); unit: U.S. Dollars ($)
Units Other Than Participants: centers
Arm/Group | Enhanced Go NAPSACC | Basic Go NAPSACC
Number analyzed (Participants) | 55 | 42
Number analyzed (centers) | 55 | 42
U.S. Dollars ($) | 154.77 (154.20) | 94.10 (143.53)

10. Secondary Outcome: Go NAPSACC Core Program Components: Percent of a TA Coaches Centers Completing Implementation Components
Description: Completion of these Go NAPSACC program components was captured using the TA activity log in Go NAPSACC website and tracking data maintained by the study interventionist and project manager. These data serve as indicators of fidelity. In the TA Activity Log all coaches document their implementation activities for each center they serve. Based on their prescribed implementation model (basic or enhanced), these data were used to calculate the percentage of a TAs centers completing the prescribed implementation activities.
Time Frame: Measures collected during the 1 year intervention period.
Population: TA coaches was the unit of analysis. For each TA coach, the percent of centers completing each outcome was computed. The TA coaches in the BASIC arm of the intervention did not have their centers: form leadership teams, complete a readiness check, or select priority areas for change. These tasks were only completed by TA coaches using the enhanced delivery model (Enhanced Go NAPSACC arm).
Measure: Number; unit: % of Centers averaged by TA coach
Units Other Than Participants: TA coaches
Arm/Group | Enhanced Go NAPSACC | Basic Go NAPSACC
Number analyzed (Participants) | 55 | 42
Number analyzed (TA coaches) | 14 | 13
% of Centers averaged by TA coach
  Registered on Go NAPSACC website | 71.4 | 85.6
  Attended Orientation meeting | 75.6 | 76.9
  Completed 9 or more Monthly Check-ins during 1 year intervention period | 19.1 | 12.2
  Formed Leadership Team: number analyzed (Participants) | 55 | 0
  Formed Leadership Team: number analyzed (TA coaches) | 14 | 0
  Formed Leadership Team | 91.7 |
  Completed Readiness check: number analyzed (Participants) | 55 | 0
  Completed Readiness check: number analyzed (TA coaches) | 14 | 0
  Completed Readiness check | 69.5 |
  Selected Priority Areas for change: number analyzed (Participants) | 55 | 0
  Selected Priority Areas for change: number analyzed (TA coaches) | 14 | 0
  Selected Priority Areas for change | 58.1 |

11. Secondary Outcome: Go NAPSACC Core Program Components: TA Coach Held Cross-Center Meetings
Description: TA coaches in the ENHANCED implementation arm were asked to hold 3 cross-center meeting during the 1 year intervention. These meeting could be online or in-person, but were intended to include directors from all centers the TA coach served. The study interventionist and project manager tracked each meeting. These data were used to calculate the percentage of prescribed implementation activities completed.
Time Frame: Measures collected during the 1 year intervention period.
Population: Cross center meetings were only completed by TA coaches (n=14) using the enhanced delivery model (Enhanced Go NAPSACC arm). The TA coaches in the BASIC arm of the intervention (n=13) did not conduct cross-center meetings. Therefore the Basic Arm is not included in analysis.
Measure: Number; unit: percent of cross-center meet held by TA
Units Other Than Participants: TA coaches
Arm/Group | Enhanced Go NAPSACC
Number analyzed (Participants) | 14
Number analyzed (TA coaches) | 14
percent of cross-center meet held by TA | 49.6

12. Secondary Outcome: Go NAPSACC Core Program Components: TA Coach Complete Logs
Description: TA coaches were asked to log implementation activities and contacts with each center in the TA Activity Log through the Go NAPSACC website. Information for analysis was extracted from the website using the TA Activity Report.
Time Frame: Measures collected during the 1 year intervention period.
Population: TA coaches who completed activity logs within Go NAPSACC website were counted as completing activity logs. TA coaches who provided no log of activities were counted as having incomplete logs.
Measure: Number; unit: percentage of TA coaches completing logs
Arm/Group | Enhanced Go NAPSACC | Basic Go NAPSACC
Number analyzed (Participants) | 14 | 13
percentage of TA coaches completing logs | 57.1 | 92.3

13. Secondary Outcome: Go NAPSACC Core Program Components: TA Coach Training Attendance
Description: TA coaches were asked to attend trainings with the study interventionist. The study interventionist and project manager tracked attendance at each training session. TA coaches in the BASIC arm were asked to attend three training sessions, while TA coaches in the ENHANCED arm were asked to attend 6 sessions. Based on their prescribed implementation model (basic or enhanced), these data were used to calculate the percentage of prescribed implementation activities completed.
Time Frame: Measures collected during the 1 year intervention period.
Population: TA coach attendance at trainings was computed and summarized over coaches in each arm.
Measure: Number; unit: percentage of trainings attended
Units Other Than Participants: TA coaches
Arm/Group | Enhanced Go NAPSACC | Basic Go NAPSACC
Number analyzed (Participants) | 14 | 13
Number analyzed (TA coaches) | 14 | 13
percentage of trainings attended | 83.3 | 96.2

14. Secondary Outcome: Go NAPSACC Core Program Components: TA Coach Attended Check-ins With Study Team
Description: TA coaches were asked to attend group check-ins with the study interventionist. The study interventionist and project manager tracked attendance at each group check-in. TA coaches in the BASIC arm were asked to attend one group check-in, while TA coaches in the ENHANCED arm were asked to attend 12 group check-ins and 3 one-on-one check-ins with study interventionist Based on their prescribed implementation model (basic or enhanced), these data were used to calculate the percentage of prescribed implementation activities completed.
Time Frame: Measures collected during the 1 year intervention period.
Population: TA coach check-in attendance was computed then summarized for each study arm.
Measure: Number; unit: percentage of check-ins attended
Units Other Than Participants: TA coaches
Arm/Group | Enhanced Go NAPSACC | Basic Go NAPSACC
Number analyzed (Participants) | 14 | 13
Number analyzed (TA coaches) | 14 | 13
percentage of check-ins attended | 83.6 | 96.2

ADVERSE EVENTS:
Time Frame: From the time of randomization through completion of the maintenance period, a total of approximately 20 months.
Description: Because adverse event reporting was collected at the person-level, sample size are based on the total number of TA coaches, directors, and staff who consented and provided data for center-level reporting.
Groups:
- Enhanced Go NAPSACC: Go NAPSACC implemented with the Enhanced delivery model,
- Basic Go NAPSACC: Go NAPSACC implemented with the Basic delivery model,
Arm/Group | Enhanced Go NAPSACC | Basic Go NAPSACC
All-Cause Mortality (participants affected / at risk) | 0/207 | 0/157
Serious Adverse Events (participants affected / at risk) | 0/207 | 0/157
Other Adverse Events (participants affected / at risk) | 0/207 | 0/157

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-01-24): https://cdn.clinicaltrials.gov/large-docs/03/NCT03938103/Prot_SAP_001.pdf
  • Informed Consent Form (2020-07-20): https://cdn.clinicaltrials.gov/large-docs/03/NCT03938103/ICF_000.pdf